CLINICAL TRIAL: NCT01736852
Title: Randomized Study to Compare the Cook Cervical Ripening Balloon (CRB) Plus Pitocin to Pitocin Alone in Premature Rupture of Membranes (PROM) Patients
Brief Title: Evaluation of CRB in PROM Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-014
Record Dates: First submitted 2012-09-06; First posted 2012-11-29 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Premature Rupture of Fetal Membranes
Keywords: Premature Rupture of Membrane (Pregnancy); PROM; Cervical Ripening; Induced Labor
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Oxytocin

ARMS (2):
- CRB plus Pitocin (Experimental)
  Interventions: Device: CRB; Drug: Pitocin
- Pitocin (Active Comparator)
  Interventions: Drug: Pitocin

INTERVENTIONS:
Device: CRB — Labor induction using the CRB
  Arms: CRB plus Pitocin
Drug: Pitocin — Labor induction using Pitocin

SUMMARY:
The CRB study is designed to study the safety and effectiveness of the Cook Cervical Ripening Balloon (CRB) for the induction of labor in term and near-term patients with premature rupture of membranes (PROM).

ELIGIBILITY:
Inclusion Criteria:

* PROM not in labor

Exclusion Criteria:

* Contraindication to vaginal delivery
* Contraindication to labor induction
* Abnormal fetal heart-rate patterns
* Maternal heart disease
* Severe maternal hypertension
* Pelvic structural abnormality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Miller, MD, Principal Investigator — Watching Over Mothers and Babies (WOMB)
Locations (4):
- United States (4):
  - Tucson Medical Center (TMC), Tucson, Arizona
  - University of South Florida, Tampa, Florida
  - Kosair Children's Hospital Maternal Fetal Medicine Specialists, Louisville, Kentucky
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request after publication of the results from this study and ending 5 years after initial publication. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CRB Plus Pitocin | Pitocin
Started | 65 | 64
Completed | 63 | 61
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRB Plus Pitocin | Pitocin | Total
Number analyzed (Participants) | 64 | 61 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (5.1) | 26.3 (5.5) | 25.7 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 61 | 125
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 2 | 5
  Black | 7 | 6 | 13
  First Nation | 5 | 2 | 7
  Hispanic or Latino | 29 | 27 | 56
  Hispanic or Latino/White | 2 | 3 | 5
  White | 18 | 21 | 39
Multiple (2 or more) previous pregnancies [Count of Participants; unit: Participants] | 31 | 28 | 59
Bishop score at time of enrollment [Mean (Standard Deviation); unit: units on a scale] — A scoring system used to assist in predicting whether induction of labor will be required. The total score is calculated by assessing the following five components on manual vaginal examination: cervical dilation, effacement, consistency, position, and fetal station. Each component is given a score of 0 to 3. The lowest possible total score would be 0 and the highest total score would be 13. The higher the total score (8 or above) the more likely a vaginal birth. The lower the score (6 or less) the more likely that intervention with a cervical ripening method may be needed to induce labor. Population: Two Patients (one in each arm) did not have their Bishop Score recorded.
  units on a scale | 4.4 (1.4) | 4.1 (1.4) | 4.2 (1.5)
Gestational age (weeks/days) [Count of Participants; unit: Participants]
  34/0 - 36/6 | 12 | 12 | 24
  37/0 - 42/6 | 52 | 49 | 101

OUTCOME MEASURES:

1. Primary Outcome: Time of Labor
Description: Time, in minutes, from the start of labor induction through delivery
Time Frame: Start of labor induction through delivery, an expected average of 6 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | CRB Plus Pitocin | Pitocin
Number analyzed (Participants) | 63 | 61
Minutes | 850.4 (417.6) | 1016.6 (595.7)

2. Primary Outcome: Incidence of Infection
Description: number of patients with chorioamnionitis
Time Frame: Through hospital discharge, an expected average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | CRB Plus Pitocin | Pitocin
Number analyzed (Participants) | 63 | 61
Participants | 7 | 6
Statistical Analysis 1: Comparison: CRB Plus Pitocin vs Pitocin; .ample size calculations were performed using an expected rate of 4% for each group,a one-sided exact test, α = 0.025, power = 0.80, non-inferiority margin of 10% resulting in a sample size of 124 patients or 62 patients per treatment arm; Test type: Non-Inferiority — non-inferiority margin of 10%, α = 0.025, power = 0.80,; p = 0.06, Fisher Exact

ADVERSE EVENTS:
Time Frame: 0-30 Days
Arm/Group | CRB Plus Pitocin | Pitocin
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/61
Serious Adverse Events (participants affected / at risk) | 5/63 | 4/61
Other Adverse Events (participants affected / at risk) | 27/63 | 21/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRB Plus Pitocin (N=63) | Pitocin (N=61)
Jaundice Neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — Hospitalization
Neonatal Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Hospitalization
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Hospitalization
Infantile Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Life Threatening
Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) — 1 Life Threatening, 1 Hospitalization
Arrested Labor (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — Hospitalization
Umbilical Cord Prolapse (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Congenital Abnormality or birth defect
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRB Plus Pitocin (N=63) | Pitocin (N=61)
Arrested Labor (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 13 (13)
Amniotic Cavity Infection (Infections and infestations) | 7 (7) | 6 (6)
Jaundice Neonatal (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications from PI prior to public release and can embargo communications of trial results between 60 and 180 days from the time submitted to the sponsor for review. The sponsor can embargo publications until the sponsor has published results or 180 days has elapsed after study closure at all participating sites. The sponsor cannot restrict publication but can require changes to protect sponsor's intellectual property rights or other confidential information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT01736852/Prot_SAP_000.pdf